CLINICAL TRIAL: NCT04486963
Title: A Randomized, Double-blind, Placebo-controlled, Ranibizumab Injected, Multicenter Phase II Clinical Study on the Efficacy and Safety of Sanhuangjingshimingwan in the Wet AMD(Qi and Yin Deficiency, Phlegm-blood Stasis Syndrome )Subjects
Brief Title: A Phase Ⅱ Clinical Study of Sanhuangjingshimingwan in Wet( Neovascular)Age-related Macular Degeneration(wAMD) Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Tasly Pharmaceutical Group Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TSL-TCM-SHJSMW-IIa
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2022-11-25 (Actual); Status verified 2022-11

CONDITIONS: Age-related Macular Degeneration
Keywords: wAMD
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sanhuangjingshimingwan group (Experimental): Sanhuangjingshimingwan,12g/bag,1 bag,Bid.Anti VEGF injection will be injected monthly if needed.
  Interventions: Drug: Sanhuangjingshimingwan
- Sanhuangjingshimingwan Placebo group (Placebo Comparator): Sanhuangjingshimingwan placebo,12g/bag,1 bag,Bid.Anti VEGF injection will be injected monthly if needed.
  Interventions: Drug: Sanhuangjingshimingwan Placebo

INTERVENTIONS:
Drug: Sanhuangjingshimingwan — Sanhuangjingshimingwan,12g,Bid,6 months.Anti VEGF injection will be injected monthly if needed.
  Arms: Sanhuangjingshimingwan group
Drug: Sanhuangjingshimingwan Placebo — Sanhuangjingshimingwan Placebo,12g,Bid,6 months.Anti VEGF injection will be injected monthly if needed.
  Arms: Sanhuangjingshimingwan Placebo group

SUMMARY:
The study is to evaluate the efficacy and safety of Sanhuangjingshimingwan in Wet AMD.

DETAILED DESCRIPTION:
The study is to evaluate the efficacy and safety of Sanhuangjingshimingwan,give two times a day versus placebo in wAMD .The clinical phase of the study comprises a 6-months double-blind treatment period, resulting in 6.5-months overall duration of the study for each patient.

ELIGIBILITY:
Inclusion Criteria:

* All patients must meet the following criteria for entry into the trail:

  1. Meet the diagnostic criteria for wAMD.
  2. Meet the Traditional Chinese Medicine diagnostic criteria for Qi and Yin Deficiency, Phlegm-blood Stasis Syndrome.
  3. Presence of choroidal neovascularization secondary to wAMD, and/or simple eye with blood, edema, leakage, hard exudation in or below the retina, and detachment of retinal pigment epithelium or neuroepithelium epithelium.
  4. 50 years≤Age≤80 years of either gender.
  5. BCVA 25 - 78 ETDRS letters(0.06~0.6, inclusive).
  6. Signed informed consent form.

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from study entry:

  1. Presence of pathological myopia,high myopia caused of secondary choroidal neovascularization, glaucoma, diabetic retinopathy, retinal arteriovenous obstruction, optic neuropathy (optic neuritis, atrophy, papillary edema), macular hole, acute phase of intraocular inflammation.
  2. Only retinal pigment epithelium-retinal detachment.
  3. The CNV area is more than 12 optic disk area (30mm2).
  4. Subfoveal structural damage or fibrosis.
  5. Subjects that have unclear refractive stroma(e.g.vitreous hemorrhage, cataracts) caused fundus observation difficulty or undergone vitrectomy.
  6. Subjects that have presence of other causes of choroidal neovascularization.
  7. Subjects that have participated in other study of treatment with study drug within the last 3 months before the screening.
  8. Subjects that have treated with photodynamic therapy, external beam radiological therapy, argon laser photocoagulation in macular area, macular surgery, transpupillary thermotherapy, hormone to treat wAMD in any eye within the last 6 months before the screening.
  9. Subjects that have undergone previous any eye surgery(except eyelid surgery).
  10. Subjects that have intravitreal anti-VEGF injections in the past 3 months.
  11. Subjects with history of fundus fluorescein and indocyanine green allergy.
  12. Subjects that have any contraindications in the directions of ranibizumab(LUCENTIS)injection.
  13. Subjects that have had severe heart disease in the last 6 months,such as congestive heart failure，unstable angina，acute coronary syndrome，myocardial infarction，Coronary revascularization，artery thrombosis, and ventricular arrhythmia that need treatment.
  14. Subjects with uncontrolled hypertension（After antihypertension treatment SBP≥140mmHg、DBP≥90mmHg）.
  15. PLT≤100×109/L; Coagulation function disorders;TBIL（Total Bilirubin）>1.5×UNL（Upper Limits of Normal）;ALT（Alanine Transaminase）>2.5×UNL or AST（Aspartate aminotransferase）>2.5×UNL;Cr（Creatinine）>1.5×UNL.
  16. Subjects with uncontrolled disease history, such as serious mental, neurological, respiratory, immune, blood and other system diseases, malignant tumors and that not suitable for the study per the investigator's judgment.

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 2020-07-24 (Actual); Primary Completion 2022-11-01 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
The average number of reinjections | at week 24
  The subject is injected with Anti-VEGF（Vascular Endothelial Growth Factor） injection once 4 weeks if needed.Compare with the average shoot number of Anti-VEGF injections in both arms.

SECONDARY OUTCOMES:
The percentage of subjects in both arms receiving reinjection of Anti-VEGF injection | at screening;at week 4;at week 8;at week 12;at week 16;at week 20;at week 24
  The subject is injected with Anti-VEGF injection once weeks if needed.Compare with the percentage of subjects who reinjected Anti-VEGF injections in both arms.
The average number of days between the second injection and baseline injection | at screening;at week 4;at week 8;at week 12;at week 16;at week 20;at week 24
  The subject is injected with Anti-VEGF injection once 4 weeks if needed.Compare with the average number of days between the second injection and baseline injection in both arms.
Change from baseline in BCVA | at screening;at week 4;at week 8;at week 12;at week 16;at week 20;at week 24
  The subject is tested the vision(BCVA) once 4 weeks with ETDRS visual chart.Compare every visit BCVA with baseline BCVA.
The BCVA increasing >5, >10 and > 15 letters change from baseline | at screening;at week 4;at week 8;at week 12;at week 16;at week 20;at week 24
  The proportion of subjects who increased BCVA >5, >10 and > 15 letters at each visit compared with the baseline.
The BCVA decreasing<5, <10 and < 15 letters change form baseline | at screening;at week 4;at week 8;at week 12;at week 16;at week 20;at week 24
  The proportion of subjects who decreased BCVA <5, <10 and <15 letters at each visit compared with the baseline.
The BCVA decreasing≥15, ≥30 letters change form baseline | at week 24
  The proportion of subjects who decreased BCVA ≥15, ≥30 letters at 24 week compared with the baseline.
Change from Baseline in Central Retinal Thickness (CRT) | at screening;at week 4;at week 8;at week 12;at week 16;at week 20;at week 24
  Change from Baseline in CRT as measured by Optical Coherence Tomography (OCT) over the study duration.
Change from Baseline in Choroidal Neovascularization (CNV) area | at screening;at week 4;at week 8;at week 12;at week 16;at week 20;at week 24
  Change from Baseline in CNV area as measured by Optical Coherence Tomography Angiography(OCTA) over the study duration.
Change from Baseline in leakage area | at week 24
  Change from Baseline in leakage area as measured by Fluorescein Angiography (FA) at week 24.
Change from Baseline in the number of polypoid choroidal vasculopathy(PCV) and Branching vascular network(BVN) area | at screening;at week 4;at week 8;at week 12;at week 16;at week 20;at week 24
  Change from Baseline in the number of PCV and BVN area as measured by Indocyanine Green Angiography(ICGA) over the study duration.
Change from Baseline in TCM(Traditional Chinese Medicine) syndrome scores | at screening;at week 4;at week 8;at week 12;at week 16;at week 20;at week 24
  The title of the scale is Traditional Chinese Medicine Syndrome Scale.Compared wth baseline,the scores of changes of TCM syndrome evaluation at each visit .This scale consists of two primary symptoms: Blurred vision and Metamorphopsia,and four secondary symptoms.Four levels to measure severity of primary symptoms（0、2、4、6）and secondary symptoms（0、1、2、3） respectively. The final score has a range of 0（none）to 42（severe）.TCM syndrome effect calculated by nimodipine method.The effect of TCM syndrome from negative (worsen) to 100% (disappear).
Change from Baseline in the effective TCM syndrome scores | at screening;at week 4;at week 8;at week 12;at week 16;at week 20;at week 24
  The title of the scale is Traditional Chinese Medicine Syndrome Scale.Compared wth baseline,the scores of changes of TCM syndrome evaluation at each visit .This scale consists of two primary symptoms: Blurred vision and Metamorphopsia,and four secondary symptoms.Four levels to measure severity of primary symptoms（0、2、4、6）and secondary symptoms（0、1、2、3） respectively. The final score has a range of 0（none）to 42（severe）.TCM syndrome effect calculated by nimodipine method.The effect of TCM syndrome from negative (worsen) to 100% (disappear).

CONTACTS AND LOCATIONS:
Overall Officials: Rui Liu, Study Director — Tasly Group, Co. Ltd.
Locations (6):
- China (6):
  - Beijing Hospital, Beijing, Beijing Municipality
  - Beijing Tongren Hospital, Beijing, Beijing Municipality
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - Shanghai General Hospital, Shanghai, Shanghai Municipality
  - Tianjin Eye Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality